CLINICAL TRIAL: NCT04354506
Title: Assessing Management of Patients With Atrial Fibrillation Through a Smart Phone Application
Brief Title: Smart Phone Atrial Fibrillation Application
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institute of Longevity (Other)
Responsible Party: Principal Investigator, Dimitris Tsiachris, Electrophysiology and Pacing Lab Director, Athens Heart Center, Institute of Longevity
Other Study IDs: AFapp
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; mobile technology
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with atrial fibrillation will have the chance to assess their disease management through an application available for free in Android and IOS smart devices

ELIGIBILITY:
Inclusion Criteria:

Paroxysmal or persistent atrial fibrillation

Exclusion Criteria:

unable to provide informed consent unable to have 1 year of follow-up for any reason

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible patients downloading specific AF mobile technology application
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | 1 year
  Clinical episodes of atrial fibrillation, hospitalisation for atrial fibrillation

SECONDARY OUTCOMES:
Stroke incidence | 1 year
  Ischemic or hemorrhagic stroke
Major bleeding incidence | 1 year
  GI bleeding, urinary bleeding necessitating hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tsiachris, MD, PHD, Study Chair — Institute of Longevity

IPD SHARING:
Plan to Share IPD: No